CLINICAL TRIAL: NCT00608946
Title: Treatment With Copper in Patients With Mild Alzheimer´s Dementia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Collaborators: University of Goettingen, Section Neurobiology (Head: Prof. Dr. T. Bayer), Germany (Other)
Responsible Party: Frank-Gerald Pajonk, M.D., Lecturer, Dept. of Psychiatry and Psychotherapy, The Saarland University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UKS-PSY-DEM-01; UKS-PSY-DEM-01
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2008-01

CONDITIONS: Alzheimer´s Disease
Keywords: efficacy of treatment with copper in patients with mild Alzheimer´s disease; cognitive status over time; CSF and volumetric data over time (1 year)
MeSH Terms: interventions — Copper

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): efficacy of the intake of 8 mg of copper daily per os for one year under observation of cognitive status unless unacceptable side effects appear
  Interventions: Dietary Supplement: copper
- 2 (Placebo Comparator): placebo
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: copper — intake of copper orotate 8 mg per day per os, once daily for one year, vs. placebo under observation of the cognitive status
  Arms: 1
Dietary Supplement: placebo — placebo
  Arms: 2

SUMMARY:
The efficacy of 8 mg of copper daily regarding cognitive function, content of beta amyloid protein in the CSF and volumetric changes in the brain will be examined in a first double-blind, placebo-controlled human clinical trial conducted in 70 patients with mild Alzheimer´s dementia.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients
* between 50 and 80 years
* criteria of mild dementia
* probable Alzheimer´s dementia according to NINCDS-ADRDA criteria
* given written informed consent
* having a relative who can fill out questionnaire; caregiver consent
* free of serious and unstable somatic illness

Exclusion Criteria:

* unable to give informed consent
* unable to take cholinesterase inhibitors
* unapproved medication
* moderate to severe Alzheimer´s disease
* dementia of other etiology
* history of alcohol, drug or medication abuse
* other psychiatric disorder, e. g. schizophrenia
* known copper and zinc storage disease
* known copper and zinc intolerance
* vegans
* known severe allergies or intolerances
* insufficient knowledge of the German language
* female patients of childbearing potential, pregnant or nursing patients
* participation in a clinical trial within the past 30 days before onset of this study
* severe somatic diseases and high mortality rate AST, ALT, GGT, GLDH, AP or bilirubin being a two-fold above the normal range

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2004-03; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
change of cognitive function, measured by ADAS-cog | one year

SECONDARY OUTCOMES:
change of beta amyloid in the CSF and volumetric changes in the brain | one year

CONTACTS AND LOCATIONS:
Overall Officials: Frank G Pajonk, M.D., lecturer, Principal Investigator — Dept. of Psychiatry and Psychotherapy, The Saarland University Hospital

REFERENCES:
- [Background] Bayer TA, Schafer S, Simons A, Kemmling A, Kamer T, Tepest R, Eckert A, Schussel K, Eikenberg O, Sturchler-Pierrat C, Abramowski D, Staufenbiel M, Multhaup G. Dietary Cu stabilizes brain superoxide dismutase 1 activity and reduces amyloid Abeta production in APP23 transgenic mice. Proc Natl Acad Sci U S A. 2003 Nov 25;100(24):14187-92. doi: 10.1073/pnas.2332818100. Epub 2003 Nov 14. PMID 14617773
- See also: Dept. of Neurobiology, University of Goettingen (Head: Prof. Dr. T. Bayer) — http://www.alzheimer-bayer.de